CLINICAL TRIAL: NCT05446493
Title: Assessment of Serum YKL-40 Level and Platelets Indices Among Patients With Diabetic Erectile Dysfunction
Brief Title: Serum YKL-40 Level and Platelets Indices Among Patients With Diabetic Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Mohamed Amer Ahmed Abdellatif, Assistant lecturer, Aswan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 346/3/19
Record Dates: First submitted 2022-01-05; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Erectile Dysfunction; Erectile Dysfunction With Diabetes Mellitus
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tadalafil group (Active Comparator): Each patient will be treated by tadalafil 5mg daily for 3months
  Interventions: Drug: Tadalafil 5mg
- control group (No Intervention): Estimation of serum YKL-40, platelet indices and serum total testosterone in healthy individuals in camparing with tadalafil group

INTERVENTIONS:
Drug: Tadalafil 5mg — * Estimate serum level of serum YKL-40, total testosterone and platelets indices in diabetic patients with erectile dysfunction treated by daily tadalafil 5mg for 3months.
  * Penile color Doppler ultrasound examination before and after treatment
  Arms: Tadalafil group

SUMMARY:
The aim of this current study is to estimate serum level of YKL-40, serum total testosterone and platelets indices in diabetic patients with erectile dysfunction treated by daily tadalafil 5mg for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with ED.

Exclusion Criteria:

* Patients with history of pelvic trauma.
* Patients with major pelvic surgical intervention.
* Patients with hypogonadism and hyperprolactinemia.
* Patients with chronic liver disease.
* Patients with cardio vascular system diseases.
* History of chronic intake of central nervous system, anti androgen drugs or other drugs as Tramadol.
* Smokers patients.
* Patients with non-vasculogenic Erectile dysfunction.

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Serum YKL-40 and platelets indices in erectile dysfunction | 3 months
  Measurement of YKL-40 and platelets indices in diabetic patients with erectile dysfunction treated by daily tadalafil.

SECONDARY OUTCOMES:
Effect of tadalafil on Erectile dysfucntion patients | 3 months
  To show the therapeutic effect of tadalafil in dose 5 mg daily on Erectile dysfucntion patients and assess their response by international index of erectile function (IIEF-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan university, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided